CLINICAL TRIAL: NCT04531891
Title: The Utility and Validity of a High-intensity, Intermittent Exercise Protocol in Male Jumping Athletes
Brief Title: Utility and Validity of a High-intensity, Intermittent Exercise Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: BC-07679
Record Dates: First submitted 2020-08-13; First posted 2020-08-31 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Each participant will randomly be assigned to two different fatigue protocols, on separate days. The first protocol is a high-intensity, intermittent exercise protocol and will be performed until complete exhaustion. The second protocol is a time-based variant of the previous protocol and will be performed during 5 minutes.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-out, high-intensity, intermittent exercise protocol (Experimental)
  Interventions: Other: Fatigue protocol
- 5 min, high-intensity, intermittent exercise protocol (Experimental)
  Interventions: Other: Fatigue protocol

INTERVENTIONS:
Other: Fatigue protocol — During the fatigue protocol, participants will sprint forward 5 m, cut at a 90° angle, sprint forward another 5 m, and backpedal 5 m. This activity will be repeated 4 times before participants will complete a series of hurdle activities. First, they will perform 2-legged jumps over 5 hurdles that are 30 cm high, turn, and repeat the jumps. Second, they will perform side-stepping exercises over the 5 hurdles. Third, they will complete four 5-m lateral shuffles.

SUMMARY:
The purpose of this study is to identify an exercise-induced fatigue protocol to mimic central and peripheral acute fatigue effects associated with participation in vigorous dynamic sports activities and to understand the expected central (cardiovascular) and peripheral (muscular) impact of this protocol.

DETAILED DESCRIPTION:
Fatigue-related parameters (BORG, heart rate, blood lactate level, concentric/eccentric force of the quadriceps muscle) will be measured before and after different short-term high-intensity, intermittent exercise protocols.

ELIGIBILITY:
Inclusion Criteria:

* Men
* ≥ 18 years
* Volley- and basketball, non-elite
* ≥ 3 times per week sports participation
* No acute or overuse low back/lower extremity injuries in the past 6 months

Exclusion Criteria:

* Women
* <18 years
* >45 years
* other sports than volley- and basketball
* elite players
* <3 times per week sports participation
* acute or overuse low back/lower extremity injuries in the past 6 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Heart rate | This parameters will be continuously monitored 10 minutes before the start of the fatigue protocol until 30 minutes after completion of the protocol
  Heart rate, expressed in beats per minute
Isokinetic dynamometry | This parameter will be monitored 10 minutes before the start of the fatigue protocol
  Isokinetic dynamometry of the quadriceps muscle
Isokinetic dynamometry | This parameter will be monitored immediately after completion of the protocol
  Isokinetic dynamometry of the quadriceps muscle
Isokinetic dynamometry | This parameter will be monitored 15 minutes after completion of the protocol
  Isokinetic dynamometry of the quadriceps muscle
Isokinetic dynamometry | This parameter will be monitored 30 minutes after completion of the protocol
  Isokinetic dynamometry of the quadriceps muscle
Blood lactate level | This parameters will be monitored 10 minutes before the start of the fatigue protocol
  Blood lactate level, expressed in millimol per liter
Blood lactate level | This parameters will be monitored 10 minutes after completion of the protocol
  Blood lactate level, expressed in millimol per liter
BORG | This parameters will be continuously monitored 10 minutes before the start of the fatigue protocol until 30 minutes after completion of the protocol
  BORG-score, indicating the rate of perceived exertion for legs and breathlessness

SECONDARY OUTCOMES:
Circuit time | Time will be recorded immediately after completion of the fatigue protocol
  Time to perform the fatigue protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep Revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
This is not yet decided.